CLINICAL TRIAL: NCT04495439
Title: Safety and Efficacy of the New ISS Sleeve Augmentation Technique in the Treatment of Osteoporotic/Osteopenic Vertebral Fractures in the Thoraco-lumbar Spine: A Pilot Study and Subsequent Comparison to the Standard PMMA-Screw Augmentation
Brief Title: Safety and Efficacy of the ISS Sleeve Augmentation Technique in the Treatment of Thoracolumbar Osteopenic Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in company strategy
Sponsor: Nexilis AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ISSCLIN-01
Record Dates: First submitted 2020-07-22; First posted 2020-07-31 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Osteoporotic Fracture of Vertebra
Keywords: bone augmentation; spine; pedicle screw; osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Polymethyl Methacrylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with ISS Sleeve (Other): The biocompatible, resorbable ISS sleeve is used for augmentation to enhance screw anchorage. It is melted into the trabecular bone structure of the osteoporotic vertebra using ultrasound. A standard pedicle screw is inserted into the sleeve.
  Interventions: Device: Augmentation with the ISS Study System
- Treatment with PMMA (Other): The bone cement Polymethylmethacrylat (PMMA) that is injected into the osteoporotic vertebra.PMMA augmentation of pedicle screws is done using standard cannulated and perforated pedicle screws. The cancellous bone surrounding the screw is enhanced with PMMA bone cement to increase screw anchorage.
  Interventions: Other: Augmentation with PMMA

INTERVENTIONS:
Device: Augmentation with the ISS Study System — Augmentation with the ISS Study System
  Arms: Treatment with ISS Sleeve
Other: Augmentation with PMMA — Augmentation with PMMA (standard)
  Arms: Treatment with PMMA

SUMMARY:
Implant anchorage is difficult in patient with osteoporotic bone. To improve the implant bone interface, the ISS stabilization system has been developed. The goal of the study is to investigate the efficacy the ISS augmentation compared to the standard PMMA augmentation of pedicle screws in the treatment of patients suffering from osteoporotic/osteopenic thoracolumbar fracture.

The study has two phases, a pilot phase followed by a pivotal phase. The data will be used to measure clinical and radiological performance and usability of both systems.

ELIGIBILITY:
Inclusion Criteria:

Patient

1. Age ≥ 50 and ≤ 85, male and female patients
2. Subject is able to understand the risks and benefits of participating in the study and is willing to provide written informed consent.
3. Psychosocially, mentally and physically able to fully comply with the protocol requirements for the duration of the study including adhering to scheduled visits, treatment plan, completing forms and other study procedures.

   Fracture
4. Fractures between the 10th thoracic and 4th lumbar vertebra, both included
5. Bone mineral density equal or above the threshold of 60 mgHA/ccm (central assessment of the screening qCT scan).
6. Fractures with the indication and possibility for augmented bi-segmental dorsal pedicle screw and rod stabilization including kyphoplasty in the broken vertebra
7. All fractures where pedicle screws can be used

Exclusion Criteria:

Patient

1. Substance use disorders (incl. tobacco abuse >20 cigarettes/day) and alcohol abuse disorders within the last 2 years before randomization.
2. BMI > 35
3. Permanent or progressive neurologic deficits (incl. upper motor neuron disease and myelopathy)
4. Known Creutzfeldt Jacob Disease
5. Systemic infections:

   * Known infection with human immunodeficiency virus (HIV) or, hepatitis B or C requiring treatment
   * Any active infection requiring the use of parenteral anti-microbial agents or that is > grade 2 Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03
6. Rheumatoid arthritis or known disorders of bone metabolism (excl. osteopenia/osteoporosis, Vitamin D deficiency)
7. Radiation therapy of the spine in medical history
8. Contraindications to pedicle screw and rod stabilization
9. Breast feeding, pregnancy or child-bearing potential (female patients of childbearing potential and male patients with a partner of child bearing potential must agree to use a highly effective contraceptive method).
10. A compromised immune system or a therapy with systemic corticosteroids or immunosuppressants
11. Active malignancy or history of malignancy (excl. Basalioma as a semi-malignant tumor) <2 years ago from time of randomization
12. Known allergy to any component of the investigational device
13. History of severe allergy, anaphylactic reactions and hypersensitivity reactions experienced in previous surgical interventions.
14. Other concurrent severe and/or uncontrolled medical conditions (e.g. insufficiently treated diabetes (HbA1c > 8 %), active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol
15. Participation in other clinical investigations for drugs or devices

    Fracture
16. Fracture age > 3 months
17. Major surgery to the spine planned for at least 12 months following enrolment
18. Any treatment of the fracture other than that specified in the inclusion criteria (e.g. index screws in the fractured vertebra, vertebroplasty, additional ventral stabilization)
19. Severe spinal deformations or fusion at the target vertebral or adjacent segments
20. Previous operations at the spine in the target or adjacent vertebrae
21. Infections or inflammatory processes at vertebral bodies

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Change of the bi-segmental kyphosis angle (Correction Loss) | Day 3 to 6 Months
  The evaluation will be done from a comparison of plain x-rays taken post-operatively before discharge (day 3 (± 1 day)) and 6 months post operatively both in upright position. The correction loss of the bi-segmental kyphosis angle will be compared in the ISS Sleeve screw augmentation group and the standard PMMA screw augmentation group.

SECONDARY OUTCOMES:
Time of x-ray exposure | Surgery
  accumulated duration; from skin incision to skin suture) of patients and medical personnel.
Compression rate | post-operatively before discharge (day 3 (± 1 day)) compared to 3, 6 and 12 months postoperatively
  Compression rate of the anterior vertebral body height measured in the lateral x-ray
Screw loosening | up to 12 months
  Screw loosening measured following the method of Aghayev et al. The angle between the axes of the pedicle screws and the cranial endplate are measured
Evaluation of the functional outcome with the Oswestry Disability | baseline, 3 months, 6 months, 12 months
  Oswestry Disability Index (ODI)
Evaluation of the pain level | baseline, 3 months, 6 months, 12 months
  Pain Scale as Visual Analogue Scale (VAS)
Evaluation of the clinical outcome | baseline, 3 months, 6 months, 12 months
  SF-12
Treatment success | at 6 and 12 months postoperatively
  composite endpoint including the correction loss of the bi-segmental kyphosis angle, the ODI and the occurrence of any device-related serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lindtner, M.D, Principal Investigator — Department of Trauma Surgery, Medical University of Innsbruck, Austria
Locations (1):
- Dept. of Orthopaedics and Traumatology, Medical University of Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No